CLINICAL TRIAL: NCT02927106
Title: Beat AML: Personalized Medicine for Acute Myeloid Leukemia Based on Functional Genomics
Brief Title: Beat AML Core Study
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Oregon Health and Science University (Other); Cellworks Group Inc. (Industry); The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Other Study IDs: IRB201601364; OCR13966 (Other: University of Florida)
Record Dates: First submitted 2016-10-05; First posted 2016-10-06 (Estimated); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Acute Myeloid Leukemia
Keywords: leukemia; myeloid; genomics
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Perform molecular and cellular studies on blood, skin biopsy, and bone marrow samples done at the time of diagnosis, after treatments, disease progression, and relapse.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Acute Myeloid Leukemia (AML): AML samples will be collected from individuals with newly diagnosed or relapsed/refractory Acute Myeloid Leukemia (AML) as defined by World Health Organization 2016.

SUMMARY:
In this study, DNA sequencing, computational biology modeling, and ex vivo drug sensitivity assays will be utilized to define clinically relevant gene mutations and identify potential therapeutics for patients with acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
As part of normal clinical care, patients will undergo a peripheral blood draw and bone marrow aspiration & biopsy. Blood draws and bone marrow aspirations are performed at the time of diagnosis, after treatments , disease progression, and relapse. Under normal clinical care, patient specimens are analyzed by cytogenetics (giemsa staining), fluorescence in situ hybridization (FISH), and gene mutation profiling. Clinically, treatment can begin before these molecular diagnostics are available.

As part of this repository study, subjects are asked to:

* Allow access to banked blood and bone marrow specimens in IRB approved protocol # 532-2012.
* Donate peripheral blood specimens whenever blood is already being drawn for clinical purposes such as at times of diagnosis, relapse, refractory disease or disease progression. Additional samples may be requested at other standard of care visits in the event that initial samples are not viable for DNA sequencing, phenotyping, or functional assays for patients with AML, if disease is present.
* Donate bone marrow aspirate specimens whenever bone marrow aspiration is already being done for clinical purposes such as at times of diagnosis, relapse, refractory disease or disease progression. If bone marrow aspirate is being collected for banking protocol #532-2012, then an aliquot of the banked specimen will be accessed rather than collect an additional bone marrow aspirate for this study.
* Undergo skin biopsy and donate the skin biopsy specimen for genomic profiling.
* Allow bone marrow, peripheral blood and skin biopsy specimens to be collected for genomic profiling and ex vivo drug sensitivity testing.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with newly diagnosed or relapsed/refractory Acute Myeloid Leukemia (AML) as defined by World Health Organization 2016.
* ≥ 18 years of age
* Capable of providing informed consent

Exclusion Criteria:

* 17 years of age or less
* greater than 80 years of age

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 50 subjects with newly diagnosed or relapsed/refractory acute myeloid leukemia (AML) will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
the genomic abnormality spectrum | 5 years
  AML cells in the peripheral blood and bone marrow samples will be examined by next generation sequencing using an Illumina DNA sequencer. DNA from the skin biopsy will be used as the constitutional reference DNA. Using skin DNA greatly improves the ability to accurately and precisely identify somatic mutations in the AML cells.
drug sensitivity | 5 years
  Ex vivo drug sensitivity testing will be performed on each subject's AML cells derived from peripheral blood and bone marrow. AML cell viability will be recorded for each treatment condition after 72 hours of treatment. A rank-ordered list of drugs will be created in order of drug toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R. Cogle, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Cancer Center, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes